CLINICAL TRIAL: NCT02583620
Title: Identification of Genomic Loci Determining Susceptibility to the Development of High Myopia
Acronym: ASSOMYP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09 036 08
Record Dates: First submitted 2015-08-18; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Myopia
Keywords: high myopia
MeSH Terms: conditions — Myopia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emmetropic volunteers (Other): Blood sample
  Interventions: Genetic: blood sample
- High myopic volunteers (Other): Blood sample
  Interventions: Genetic: blood sample

INTERVENTIONS:
Genetic: blood sample — A blood test is realized on the subject

SUMMARY:
Compelling evidence of genetic components in high myopia has been put forward by several studies. Twin cohorts, familial linkage studies and population studies has described at least 10 loci containing genes involved in the disease development. The investigators previously demonstrated novel linkage on chromosome 7q36 and chromosome 7p15 in French families. A new approach consisting of a case-control based population association study is underway in order to recover a high number of myopic subjects avoiding the limitation of familial cases. 1.8 millions polymorphic markers will be compared with emmetropic controls in order to recover loci associated with the disease in the population.

DETAILED DESCRIPTION:
Myopia is a worldwide refractive ocular disorder and is the most frequent visual defect in man. It is responsible for a major health problem, affecting around 25% of the western population. High myopia is the most severe form of the myopic spectrum and is defined by an increase of refractive error beyond -5 dioptres. About 2.5% of the general population suffers from this, while the secondary complications are responsible among these patients for the 4th cause of legal blindness. The physiopathology of myopia remains unknown and mechanisms leading to the disease are most probably complex, mixing acquired environmental and genetics factors. Our team in a previous study gathered and analysed an important series of high myopic families: Heritability, segregation and linkage analyses modelling the transmission mode localised two major genomic regions linked to high myopia susceptibility on chromosome 7q36 and chromosome 7p15. Several loci have been described by other teams working on the same topic among different human populations. Very recently reappraisal of 55 families led to the delineation of a complex segregation model of the high myopia phenotype thus claiming an oligo- polygenic mode of transmission. Together these results express the need to collect more cases and to substitute an linkage studies by association studies already conducted in order to increase the power to detect involved loci.

To find one or more genomic loci involved in high myopia susceptibility; a polygenic model and association analysis is considered a referent method to decipher the participation of multiple, low acting loci. High density SNPs/CNVs DNA markers covering the whole genome will be used for genotyping.

Phenotypes including ophthalmologic evaluation, ethno-geographic origin and familial data will be collected in order to allow further stratification or clustering.

Computing of the statistical power of the association analysis conducted to minimize the number of false positive associations and to obtain a 80% of detection power indicated the need of 400 high myopic subjects and 400 controls to be analysed.

Collaboration between a Clinical Investigation Center (CIC) and Ophthalmology clinics will be used to overcome recruitment problems. DNA extraction and genotyping will be conducted in Institut national de la santé et de la recherche (INSERM-UPS) unit in Toulouse using the "Toulouse's Génopole" microarrays genotyping facilities.

ELIGIBILITY:
Inclusion Criteria:

* high myopic (cases) volunteers,
* emmetropic (controls) volunteers

Exclusion Criteria:

* syndromic myopic children under 18 years,
* non autonomous adults

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2009-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Numbers of allele frequencies at markers in the population | Baseline
  Numbers of allele frequencies at markers in the population

CONTACTS AND LOCATIONS:
Overall Officials: François MALECAZE, PhD, MD, Principal Investigator — University Hospital, Toulouse
Locations (4):
- France (4):
  - CHU Pointe-à-Pitre, Pointe à Pitre, Guadeloupe
  - CHU Bordeaux Hôpital Pellegrin, Bordeaux
  - CHU Limoges Hôpital Dupuytren, Limoges
  - CHU Toulouse Hôpital Purpan, Toulouse